CLINICAL TRIAL: NCT03407820
Title: Randomized Controlled Trial Comparing Nylon and Chromic Gut Sutures After Minor Hand Surgery
Brief Title: Nylon Versus Chromic Gut Sutures for Minor Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, Associate Dean for Comprehensive Care. Professor of Surgery and Psychiatry, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-11-0021
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: All Minor Hand Surgery Including; Carpal Tunnel Syndrome; Trigger Finger; Ganglion Cysts; De Quervain Syndrome; Dupuytren Contracture
MeSH Terms: conditions — Carpal Tunnel Syndrome; Trigger Finger Disorder; Ganglion Cysts; Dupuytren Contracture

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Both patient and surgeon will be blinded until just before the start of the procedure.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st random 50% of cohort (Active Comparator): Absorbable Chromic gut sutures
  Interventions: Procedure: Absorbable Chromic gut sutures
- 2nd random 50% of cohort (Active Comparator): Non-absorbable Nylon sutures
  Interventions: Procedure: Non-absorbable Nylon sutures

INTERVENTIONS:
Procedure: Absorbable Chromic gut sutures — In this group interrupted simple or horizontal mattress skin sutures are used for wound closure per surgeon preference. Standardized wound care instructions will be given to all patients. Those who received absorbable Chromic sutures are treated recording to the standard protocol and they are advised that they can start to gently rub the scab and suture line to encourage the sutures to fall off starting 10-14 days postoperatively.
  Arms: 1st random 50% of cohort
Procedure: Non-absorbable Nylon sutures — In this group interrupted simple or horizontal mattress skin sutures are used for wound closure per surgeon preference. Standardized wound care instructions will be given to all patients. Those who received Nylon sutures are treated recording to the standard protocol and sutures are removed after the usual time (10-14 days) of the received procedure.
  Arms: 2nd random 50% of cohort

SUMMARY:
This study aims to assess the relationship between overall satisfaction with treatment in a group of randomized patients undergoing elective hand surgery using either absorbable (4-0 Chromic) or non-absorbable (5-0 Nylon) sutures. The investigators will also assess factors associated with wound concerns, pain intensity, magnitude of limitations, and physical function within one month of surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing common day-case elective hand surgery under local anesthesia, one of the following (initial) procedures:

  * Carpal tunnel release
  * Trigger finger release
  * Ganglion excision
  * Excisional biopsy
  * De Quervain release
  * Dupuytren fasciectomy
  * Any other minor hand surgery
* Patients aged 18-89
* Able to provide informed consent
* Able to understand English or Spanish to complete questionnaires
* Patients who have an email-address or phone number (needed for follow-up)
* UT Health Austin Musculoskeletal Institute, Austin Regional Clinic, Orthopaedic Specialists of Austin.
* Available for follow-up contact after 4 weeks

Exclusion Criteria:

* Patients not able to give informed consent
* Patients using corticosteroids
* Patients with one of the following comorbidities: bleeding disorder, immunodeficiency, collagen vascular disease.
* Patients known to be allergic to suture materials
* Revision procedures

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Treatment satisfaction measured on an 11-point ordinal scale | Four weeks after surgery
  The scale ranges from 0 to 10, with higher scores representing higher treatment satisfaction.

SECONDARY OUTCOMES:
Factors associated with wound concerns within one month of surgery | Four weeks after surgery
  Factors will include patient demographic factors such as age, sex, race/ethnicity, level of education. Wound concerns will be assessed by number of contacts with questions for wound concerns.
Factors associated with pain intensity (11 point ordinal scale) within one month of surgery | Four weeks after surgery
  Factors will include patient demographic factors such as age, sex, race/ethnicity, level of education. The scale ranges from 0 to 10, with higher scores representing higher pain intensity.
Factors associated with magnitude of limitations (with PROMIS-UE PF) within one month of surgery | Four weeks after surgery
  Factors will include patient demographic factors such as age, sex, race/ethnicity, level of education. PROMIS-UE PF scores are reported as T-scores with a mean of 50 and SD of 10, with higher scores representing higher levels of physical function.
Factors associated with scar satisfaction (11 point ordinal scale) within one month of surgery | Four weeks after surgery
  Factors will include patient demographic factors such as age, sex, race/ethnicity, level of education. The scale ranges from 0 to 10, with higher scores representing higher scar satisfaction.
Difference in treatment satisfaction between patients rating 0-8 and 9-10 on an 11-point ordinal scale | Four weeks after surgery
  he scale ranges from 0 to 10, with higher scores representing higher treatment satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD PhD, Principal Investigator — University of Texas at Austin
Locations (3):
- United States (3):
  - Austin Regional Clinic, Austin, Texas
  - HTB Musculoskeletal Institute, Austin, Texas
  - Orthopedic Specialists of Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: No